CLINICAL TRIAL: NCT00270166
Title: A Placebo-Controlled Study on the Effect of Epoetin Alfa in Patients With Malignancy Receiving Chemotherapy
Brief Title: The Effect of Epoetin Alfa on the Anemia of Patients With Selected Cancers Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005923
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-02

CONDITIONS: Anemia; Multiple Myeloma; Lymphoma; Breast Cancer; Ovarian Cancer; Carcinoma, Small Cell Lung; Esophagus Cancer; Prostate Cancer; Neoplasm
Keywords: cancer; malignancy; red cell transfusion; epoetin alfa; epoetin; erythropoietin; red blood cells
MeSH Terms: conditions — Anemia; Multiple Myeloma; Lymphoma; Breast Neoplasms; Ovarian Neoplasms; Small Cell Lung Carcinoma; Esophageal Neoplasms; Prostatic Neoplasms; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa versus placebo in reducing or preventing the need for transfusions in anemic patients with cancer receiving chemotherapy, and to investigate possible quality-of-life benefits associated with the use of epoetin alfa. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy, or both. Quality of life is also affected, in part because of the fatigue associated with anemia. Previous studies with epoetin alfa have suggested that achieving a higher hemoglobin level may improve quality of life and help patients live longer. This study is a 12-week, double-blind, placebo-controlled multicenter study to compare the ability of epoetin alfa and placebo in reducing or preventing anemia and transfusions, and to investigate quality-of-life benefits associated with the use of epoetin alfa in patients receiving chemotherapy for selected cancers. During the double-blind period there will be two groups of patients: one group receiving epoetin injections under the skin 3 times per week (starting at 150 units per kilogram, adjusted if needed to a maximum of 300 units per kilogram) and other group receiving injections under the skin of a placebo of matching appearance and volume. If hemoglobin rises above 140 grams per liter (women) or 150 grams per liter (men), the dose will be adjusted to keep hemoglobin within a target range. A 12-week open-label extension of the study will be available to all patients completing the 12-week comparison period. The primary measure of effectiveness is determined by the proportion of patients with no transfusions after the first month. Additional measures of effectiveness include: the proportion of responders, the change of hemoglobin unrelated to transfusion, cumulative transfusion rate and proportion of patients transfused during the double-blind phase (excluding the first month), as well as the mean change over the study period in scores for energy, activity and overall quality of life. The results will be analyzed separately for non-platinum-containing chemotherapy and for different tumor types. Safety evaluations include assessments of the incidence and severity of adverse events, clinical laboratory tests, vital sign measurements, and physical examinations. The hypothesis of the study is that epoetin alfa is superior to placebo in improving anemia, reducing the number of transfusions, and improving quality of life. Epoetin alfa 150 units (U) per kilogram (kg) or placebo, injected under the skin 3 times weekly for 4 weeks; then either continued at 150 U/kg or adjusted to 300 U/kg according to hemoglobin levels for the remaining 8 weeks. Open-label (12 weeks): dose to maintain target hemoglobin range.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma, lymphoma, breast cancer, ovarian cancer, small-cell lung cancer, esophagus cancer, or prostate cancer
* receiving treatment with chemotherapy, with at least 3 additional months of chemotherapy planned
* a self-care performance score of 0 (fully active, no disease restriction) to 3 (capable of only limited self-care, confined to bed or chair more than 50% of waking hours)
* life expectancy of at least 6 months
* baseline hemoglobin <12 grams per deciliter and baseline count of <100,000 microliter for developing red cells

Exclusion Criteria:

* Clinically significant disease other than cancer
* evidence of uncontrolled hypertension or history of seizure
* transfusion within 1 week of the study
* radiotherapy within 2 weeks of study start
* use of corticosteroid or steroid drugs during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 1995-02; Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without transfusion after first month.

SECONDARY OUTCOMES:
Proportion of responders, change of hemoglobin (not by transfusion), cumulative transfusion rate, proportion of patients transfused during the double-blind phase, excluding the first month; mean change score of baseline quality of life parameters; safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: The effect of epoetin alfa on the anemia of patients with selected cancers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=686&filename=CR005923_CSR.pdf